CLINICAL TRIAL: NCT02866266
Title: Extended Release (ER) / Long-acting (LA) Opioid Analgesics Risk Evaluation and Mitigation Strategy (REMS) Assessment 5.1: Surveillance of Emergency Department Visits and Hospitalizations for Opioid Overdose and Poisoning Events
Brief Title: ER/LA Opioid Surveillance for Emergency Department Visits and Hospitalizations for Overdose and Poisoning
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ER/LA Opioid REMS Program Companies (RPC) (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Assessment 5.1
Record Dates: First submitted 2016-06-08; First posted 2016-08-15 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Opioid-related Disorders; Opioid Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- All commercially insured patients in the HIRD
  Interventions: Other: Retrospective database review
- All Medicaid patients in a participating state Medicaid plan
  Interventions: Other: Retrospective database review

INTERVENTIONS:
Other: Retrospective database review

SUMMARY:
Study to evaluate the impact of the ER/LA opioid REMS program on the incidence of Emergency Department visits and hospitalizations for overdose/poisoning and death among patients prescribed ER/LA opioid analgesics.

DETAILED DESCRIPTION:
As part of the FDA-approved plan to evaluate the effects of the REMS program, the REMS Program Companies (RPC) are required to submit FDA assessment reports on a regular basis. The present study is one of several program evaluation components carried out in support Assessment 5: Surveillance monitoring for misuse, abuse, overdose, addiction, death and intervention taken. This study will evaluate the impact of the ER/LA opioid REMS program on the incidence of ED visits and hospitalizations for overdose/poisoning and death among patients prescribed ER/LA opioid analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. At least one dispensing of an ER/LA opioid after 01 July 2010
2. At least six months of continuous health plan eligibility prior to the first recorded dispensing of an opioid that occurs during an included REMS period

Exclusion Criteria:

1. Missing or implausible values for age
2. Missing or implausible values for gender

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients that receive at least one dispensing of an ER/LA opioid during at least one study REMS period with at least six months of prior continuous health plan eligibility in the main analyses. Additional analyses will consider patients enrolled in the HIRD or a participating Medicaid plan regardless of ER/LA opioid exposure.
Sampling Method: Non-Probability Sample
Enrollment: 183452 (Actual)
Dates: Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of ED visits for opioid overdose/poisoning and mortality | Retrospective review over period from July 2010 through December 2014
Number of hospitalizations for opioid overdose/poisoning and mortality | Retrospective review over period from July 2010 through December 2014

SECONDARY OUTCOMES:
All-cause mortality | Retrospective review over period from July 2010 through December 2014